CLINICAL TRIAL: NCT02570815
Title: Near-Infrared Fluorescence Guided Robotic Pulmonary Segmentectomy for Early Stage Lung Cancer: Analysis of Accuracy and Added Value
Brief Title: Near-Infrared Fluorescence Guided Robotic Pulmonary Segmentectomy for Early Stage Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Wael Hanna, Director, Research Program, Boris Family Centre for Robotic Surgery, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFCRS-RP-001-1504-29; 101 (Other: Hamilton Integrated Research Ethics Board)
Record Dates: First submitted 2015-09-22; First posted 2015-10-07 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: lung cancer; segmentectomy; robotic surgery; near-infrared fluorescent; IC-GREEN; indocyanine green; early-stage lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- indocyanine green (Experimental): Non-toxic, fluorescent dye
  Interventions: Drug: indocyanine green

INTERVENTIONS:
Drug: indocyanine green — ICG will be prepared as a sterile solution (2.5 mg/10mL) for injection. After vascular ligation, a 6 to 8mL bolus of ICG solution will be injected into the peripheral vein catheter, followed by a 10mL saline solution bolus. The Firefly camera will then be used for the NIF imaging. It is expected that the entire lung, except the segment which was previously isolated from blood supply, will fluoresce within 30-40 seconds, exhibiting a green hue. The surgeon will perform the pulmonary resection and the resected 'dark' lung segment will be immediately evaluated by a pathologist, depending on the pathologist findings the operation may be concluded or the patient will receive a pulmonary lobectomy.
  Other Names: IC-GREEN

SUMMARY:
Lungs are made up of individual lobes. When a lung cancer tumour is detected in one of these lobes, surgeons typically perform a Lobectomy. A Lobectomy is the surgery most commonly done to treat early-stage lung cancer and requires removal of an entire lobe of the lung, which removes a large amount of lung tissue For patients with small tumours saving as much healthy lung tissue as possible is important. Each lobe of the lung has smaller sections called segments. When a lung cancer is in one of these segments, it is possible to remove that segment, without removing the entire lobe. This surgery is called a segmentectomy. Compared to a lobectomy, a segmentectomy saves a larger amount of healthy lung tissue.

With the advances in screening technology for lung cancer tumours, an increasing amount of very small lung cancer tumours are being found, and the demand for segmentectomy is increasing. A segmentectomy is a hard surgery to perform robotically because it is difficult to view the tissue lines that separate each segment within the lobe. As a result, it is difficult for the surgeon to see exactly which pieces of tissue should be removed. Because of these challenges, many patients having robotic surgery will have a lobectomy, even if a full lobectomy is not needed.

Near-Infrared Fluorescence (NIF) using indocyanine green (ICG) fluorescent dye is a recent advancement in the robotic platform of robotic surgery. The surgeon will view the CT scan to determine which segment the tumour is located in. Once identified, the surgeon will isolate the segment by cutting off the blood supply to that segment. Then ICG will be injected into a vein. It is expected that the entire lung, except the isolated segment, which will remain 'dark' as it was isolated from blood supply, will fluoresce, giving off a green hue when viewed with the da Vinci Firefly camera. The surgeon will identify 'dark' segment, and will remove it. A pathologist will examine the excised tissue to ensure that the tumour was removed in its entirety. Once confirmed, the surgeon will end the procedure. If the pathologist determines that the segment removed did not contain the entire tumour, then the surgeon will perform a routine lobectomy. This ensures patient safety and confirms that all participants will have the entire tumour removed from their lung.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Tumor size <3 cm
3. Clinical Stage 1 Non-Small Cell Lung Cancer (NSCLC)
4. CT-imaging confirming that the tumour is confined to the one broncho-pulmonary segment, rendering the patient a candidate for segmental resection.

Exclusion Criteria:

1. Hypersensitivity or allergy to ICG, sodium iodide or iodine
2. Women who are currently pregnant or are breast feeding; or women of child bearing potential who are not currently taking adequate birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-10; Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using NIF-guidance in robotic pulmonary segmentectomy for early-stage lung cancer will be evaluated using items 1, 2, and 3 of a 7-item binary rating scale. An score of 3/7 for these items will indicate success. | 1 year
  Item 1: Visualization of fluoresced lung by NIF imaging; Item 2:Demarcation of a dark segment and inter-segmental plane; Item 3: Completion of segmental resection along the borders of the dark-segmental plane.

SECONDARY OUTCOMES:
Safety will be measured by the rate of adverse reactions to ICG dye as defined by the Ottawa Thoracic Morbidity and Mortality classification | 1 year
Safety will also be measured by the rate of perioperative complications as defined by the Ottawa Thoracic Morbidity and Mortality classification | 1 year
Anatomical accuracy will be evaluated using items 4, 5, and 6 of the Indocyanine Green Segmentectomy 7-Item Binary Scale. A score of 3/7 on these items will indicate success of anatomical accuracy | 1 year
  Item 4: Ex-vivo localization of lesions; Item 5: Ex-vivo confirmation of tumor-free margins around lesion; Item 6: Ex-vivo confirmation of adequate anatomical inter-segmental.
Added value of ICG-guidance will be evaluated using Item 7 of the 7-item binary rating scale. A score of 1/7 will indicate added value of ICG-guidance | 1 year
  Item 7: Added value of NIF-guidance
Overall success of the intervention will be evaluated using Items 1-7 of the binary rating scale, only an aggregate score of 7/7 will be considered a success | 1 year
Reproducibility and validity of the procedure will be measured by the rate of overall success | 1 year
Partial success of the intervention will be measured by scores between 1/5 and 4/5 on the 7-item binary scale | 1 year
Length of time of the procedure will be measured by collecting the procedure start and procedure start time | 1 year
Length of time of the operation will be measured by collecting the time the patient entered the operating room until the time the patient left the operating room | 1 year
Rate of conversions to lobectomy will be measured by collecting the proportion of conversions to lobectomy or thoracotomy | 1 year
Rate of conversion to thoracotomy will be measured by collecting the proportion of conversions to thoracotomy | 1 year
Duration the patient had chest tubes in situ will be measured by collecting the date of surgery and the date the chest tube was removed | 1 year
Duration of hospital length of stay will be measured by collecting the data of admission and the date of discharge | 1 year
Learning Curve | 1 year
  Learning curve will be evaluated during the analysis of the data using Items 1-7 of the 7-item binary rating scale, particularly the measured difference (millimeters) in the predicted cautery-marked intersegmental planes delineated prior to using ICG and the true anatomical intersegmental planes delineated with ICG and NIF.

CONTACTS AND LOCATIONS:
Overall Officials: Waël C. Hanna, MDCM, MBA, FRCSC, Principal Investigator — St. Joseph's Healthcare Hamilton / McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Landreneau RJ, Sugarbaker DJ, Mack MJ, Hazelrigg SR, Luketich JD, Fetterman L, Liptay MJ, Bartley S, Boley TM, Keenan RJ, Ferson PF, Weyant RJ, Naunheim KS. Wedge resection versus lobectomy for stage I (T1 N0 M0) non-small-cell lung cancer. J Thorac Cardiovasc Surg. 1997 Apr;113(4):691-8; discussion 698-700. doi: 10.1016/S0022-5223(97)70226-5. PMID 9104978
- [Background] Zhao X, Qian L, Luo Q, Huang J. Segmentectomy as a safe and equally effective surgical option under complete video-assisted thoracic surgery for patients of stage I non-small cell lung cancer. J Cardiothorac Surg. 2013 Apr 29;8:116. doi: 10.1186/1749-8090-8-116. PMID 23628209
- [Background] Pardolesi A, Veronesi G, Solli P, Spaggiari L. Use of indocyanine green to facilitate intersegmental plane identification during robotic anatomic segmentectomy. J Thorac Cardiovasc Surg. 2014 Aug;148(2):737-8. doi: 10.1016/j.jtcvs.2014.03.001. Epub 2014 Mar 5. No abstract available. PMID 24680390
- [Background] Finley RJ, Mayo JR, Grant K, Clifton JC, English J, Leo J, Lam S. Preoperative computed tomography-guided microcoil localization of small peripheral pulmonary nodules: a prospective randomized controlled trial. J Thorac Cardiovasc Surg. 2015 Jan;149(1):26-31. doi: 10.1016/j.jtcvs.2014.08.055. Epub 2014 Sep 16. PMID 25293355
- [Background] Ivanovic J, Al-Hussaini A, Al-Shehab D, Threader J, Villeneuve PJ, Ramsay T, Maziak DE, Gilbert S, Shamji FM, Sundaresan RS, Seely AJ. Evaluating the reliability and reproducibility of the Ottawa Thoracic Morbidity and Mortality classification system. Ann Thorac Surg. 2011 Feb;91(2):387-93. doi: 10.1016/j.athoracsur.2010.10.035. PMID 21256276